CLINICAL TRIAL: NCT02617810
Title: An Open-Label Drug Interaction Study to Assess the Effect of Multiple-Dose Administration of JNJ-42847922 on the Single-Dose Pharmacokinetics of Midazolam and the Single Dose Pharmacokinetics and Pharmacodynamics of Warfarin in Healthy Subjects
Brief Title: A Study to Assess the Effect of Multiple-Dose Administration of JNJ-42847922 on Midazolam and Warfarin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108066; 42847922EDI1010 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-11-13; First posted 2015-12-01 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
Keywords: Healthy; JNJ-42847922; Midazolam; Warfarin; Pharmacokinetics
MeSH Terms: interventions — seltorexant; Midazolam; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- JNJ-42847922 Plus Midazolam Plus Warfarin (Experimental): Participants will receive Treatment A (midazolam 4 milligram [mg] syrup once on Day 1 and warfarin 25 mg tablet once on Day 3) followed by Treatment B (JNJ-42847922 20 mg once daily from Day 1 to Day 9, midazolam 4 mg syrup once on Day 7 and warfarin 25 mg tablet once on Day 9). A washout period of 14 to 21 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-42847922; Drug: Midazolam; Drug: Warfarin

INTERVENTIONS:
Drug: JNJ-42847922 — Participants will receive JNJ-42847922 20 milligram (mg) tablet orally once daily from Day 1 to Day 9.
Drug: Midazolam — Participants will receive midazolam 4 milligram (mg) syrup orally once on Day 1 during treatment A and on Day 7 during treatment B.
Drug: Warfarin — Participants will receive warfarin 25 milligram (mg) tablet orally once on Day 3 during treatment A and on Day 9 during treatment B.

SUMMARY:
The purpose of this study is to evaluate effect of multiple-dose administration of JNJ-42847922 on the single-dose pharmacokinetics of oral midazolam and single-dose pharmacokinetics and pharmacodynamics of (R)- and (S)-warfarin after oral administration of racemic warfarin.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single-center, fixed-sequence, study of JNJ-42847922 in healthy participants. The study consists of 3 Phases: Screening Phase (28 Days), open-label treatment Phase (40 Days) and follow up visit (7 to 14 Days after last study procedure). The duration of participation in the study for each participant is approximately 82 Days. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study
* Willing to adhere to the prohibitions and restrictions specified in protocol
* If a woman, must be not of child-bearing potential: postmenopausal [greater than or equal to (>=) 45 years of age with amenorrhea for at least 2 years, or any age with amenorrhea for at least 6 months and a serum stimulating hormone (FSH) greater than (>) 40 International units per liter (IU/L), or surgically sterile (example, hysterectomy, oophorectomy, tubal ligation or tubal occlusion)
* If a woman, must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction for at least 3 months after the last dose of study drug
* If a man who is sexually active with a woman of childbearing potential and has not had a vasectomy, must agree to use an adequate contraception method as deemed appropriate by the Investigator (example, vasectomy, double-barrier, partner using effective contraception) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Body mass index (BMI) between 18 and 30 kilogram (kg)/meter^2 (m^2), and body weight not less than 50 kg

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), syncope, hypotension, hypertension or vascular disorders, lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, kidney or urinary tract disturbances, thyroid disease, neurologic disease, significant psychiatric disorder, epilepsy, or fits of unexplained black-outs, infection, or any other illness that the Investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry, urinalysis, or thyroid stimulating hormone (TSH) at Screening or at Day -1 of the first treatment period as deemed appropriate by the Investigator. In addition, participants must have coagulation test results [(prothrombin time (PT), international normalized ratio (INR), and activated partial thromboplastin time (aPTT)] within clinically acceptable limits at Screening as deemed appropriate by the Investigator
* Clinically significant abnormal physical examination, vital signs, or 12 lead electrocardiogram (ECG) at Screening or Day -1 of the first treatment period as deemed appropriate by the Investigator
* Participants who are homozygous or heterozygous for CYP2C9*2 or CYP2C9*3 alleles
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for acetaminophen, within 14 days before the first dose of the study drug is scheduled until completion of the study. In addition, participants will be excluded if they have used medications known to affect coagulation or modulate CYP2C9 or VKORC1 within 28 days of study admission

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Midazolam | Predose, 0.5, 1, 1.5, 2, 3 , 4, 6, 8, 10, 12, 16, 24, 30, 36 and 48 hours postdose on Day 1 during Treatment A and on Day 7 during Treatment B
  The Cmax is the maximum observed plasma concentration of Midazolam.
Maximum Plasma Concentration (Cmax) of 1-Hydroxymidazolam | Predose, 0.5, 1, 1.5, 2, 3 , 4, 6, 8, 10, 12, 16, 24, 30, 36 and 48 hours postdose on Day 1 during Treatment A and on Day 7 during Treatment B
  The Cmax is the maximum observed plasma concentration of 1-Hydroxymidazolam.
Maximum Plasma Concentration (Cmax) of Warfarin | Predose, 0.5, 1, 2 , 4, 6, 9, 12, 16, 24, 36, 48, 72, 96, 120, 144 and 168 hours postdose on Day 3 during Treatment A and on Day 9 during Treatment B
  The Cmax is the maximum observed plasma concentration of Warfarin.
Time to Reach the Maximum Plasma Concentration (Tmax) of Midazolam | Predose, 0.5, 1, 1.5, 2, 3 , 4, 6, 8, 10, 12, 16, 24, 30, 36 and 48 hours postdose on Day 1 during Treatment A and on Day 7 during Treatment B
  The Tmax is the time to reach the maximum observed plasma concentration of Midazolam.
Time to Reach the Maximum Plasma Concentration (Tmax) of 1-Hydroxymidazolam | Predose, 0.5, 1, 1.5, 2, 3 , 4, 6, 8, 10, 12, 16, 24, 30, 36 and 48 hours postdose on Day 1 during Treatment A and on Day 7 during Treatment B
  The Tmax is the time to reach the maximum observed plasma concentration of 1-Hydroxymidazolam.
Time to Reach the Maximum Plasma Concentration (Tmax) of Warfarin | Predose, 0.5, 1, 2 , 4, 6, 9, 12, 16, 24, 36, 48, 72, 96, 120, 144 and 168 hours postdose on Day 3 during Treatment A and on Day 9 during Treatment B
  The Tmax is the time to reach the maximum observed plasma concentration of Warfarin.
Time of Last Measurable Plasma Concentration (Tlast) of Midazolam | Predose, 0.5, 1, 1.5, 2, 3 , 4, 6, 8, 10, 12, 16, 24, 30, 36 and 48 hours postdose on Day 1 during Treatment A and on Day 7 during Treatment B
  Time to last measurable plasma concentration is evaluated.
Time of Last Measurable Plasma Concentration (Tlast) of 1-Hydroxymidazolam | Predose, 0.5, 1, 1.5, 2, 3 , 4, 6, 8, 10, 12, 16, 24, 30, 36 and 48 hours postdose on Day 1 during Treatment A and on Day 7 during Treatment B
  Time to last measurable plasma concentration is evaluated.
Time of Last Measurable Plasma Concentration (Tlast) of Warfarin | Predose, 0.5, 1, 2 , 4, 6, 9, 12, 16, 24, 36, 48, 72, 96, 120, 144 and 168 hours postdose on Day 3 during Treatment A and on Day 9 during Treatment B
  Time to last measurable plasma concentration is evaluated.
Area Under the Plasma Concentration-Time Curve From 0 to Last Quantifiable Concentration (AUC[0-last]) Post Dose of Midazolam | Predose, 0.5, 1, 1.5, 2, 3 , 4, 6, 8, 10, 12, 16, 24, 30, 36 and 48 hours postdose on Day 1 during Treatment A and on Day 7 during Treatment B
  The AUC(0-last) is the area under the plasma concentration-time curve from 0 to time of the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From 0 to Last Quantifiable Concentration (AUC[0-last]) Post Dose of 1-Hydroxymidazolam | Predose, 0.5, 1, 1.5, 2, 3 , 4, 6, 8, 10, 12, 16, 24, 30, 36 and 48 hours postdose on Day 1 during Treatment A and on Day 7 during Treatment B
  The AUC(0-last) is the area under the plasma concentration-time curve from 0 to time of the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From 0 to Last Quantifiable Concentration (AUC[0-last]) Post Dose of Warfarin | Predose, 0.5, 1, 2 , 4, 6, 9, 12, 16, 24, 36, 48, 72, 96, 120, 144 and 168 hours postdose on Day 3 during Treatment A and on Day 9 during Treatment B
  The AUC(0-last) is the area under the plasma concentration-time curve from 0 to time of the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From 0 to Infinite Time (AUC[0-infinity]) Post Dose of Midazolam | Predose, 0.5, 1, 1.5, 2, 3 , 4, 6, 8, 10, 12, 16, 24, 30, 36 and 48 hours postdose on Day 1 during Treatment A and on Day 7 during Treatment B
  The AUC (0-infinity) is the area under the plasma Midazolam concentration-time curve from time 0 to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z), in which AUC(0-last) is area under the plasma Midazolam concentration-time curve from time zero to time of the last quantifiable concentration, C(last) is the last observed quantifiable concentration and lambda(z) is elimination rate constant.
Area Under the Plasma Concentration-Time Curve From 0 to Infinite Time (AUC[0-infinity]) Post Dose of 1-Hydroxymidazolam | Predose, 0.5, 1, 1.5, 2, 3 , 4, 6, 8, 10, 12, 16, 24, 30, 36 and 48 hours postdose on Day 1 during Treatment A and on Day 7 during Treatment B
  The AUC (0-infinity) is the area under the plasma 1-Hydroxymidazolam concentration-time curve from time 0 to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z), in which AUC(0-last) is area under the plasma 1-Hydroxymidazolam concentration-time curve from time zero to time of the last quantifiable concentration, C(last) is the last observed quantifiable concentration and lambda(z) is elimination rate constant.
Area Under the Plasma Concentration-Time Curve From 0 to Infinite Time (AUC[0-infinity]) Post Dose of Warfarin | Predose, 0.5, 1, 2 , 4, 6, 9, 12, 16, 24, 36, 48, 72, 96, 120, 144 and 168 hours postdose on Day 3 during Treatment A and on Day 9 during Treatment B
  The AUC (0-infinity) is the area under the plasma Warfarin concentration-time curve from time 0 to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z), in which AUC(0-last) is area under the plasma Warfarin concentration-time curve from time zero to time of the last quantifiable concentration, C(last) is the last observed quantifiable concentration and lambda(z) is elimination rate constant.
Terminal Half-life (t[1/2]) of Midazolam | Predose, 0.5, 1, 1.5, 2, 3 , 4, 6, 8, 10, 12, 16, 24, 30, 36 and 48 hours postdose on Day 1 during Treatment A and on Day 7 during Treatment B
  Elimination half-life associated with the terminal slope Lambda (z) of the semi logarithmic drug concentration-time curve, calculated as 0.693/Lambda (z).
Terminal Half-life (t[1/2]) of 1-Hydroxymidazolam | Predose, 0.5, 1, 1.5, 2, 3 , 4, 6, 8, 10, 12, 16, 24, 30, 36 and 48 hours postdose on Day 1 during Treatment A and on Day 7 during Treatment B
  Elimination half-life associated with the terminal slope Lambda (z) of the semi logarithmic drug concentration-time curve, calculated as 0.693/Lambda (z).
Terminal Half-life (t[1/2]) of Warfarin | Predose, 0.5, 1, 2 , 4, 6, 9, 12, 16, 24, 36, 48, 72, 96, 120, 144 and 168 hours postdose on Day 3 during Treatment A and on Day 9 during Treatment B
  Elimination half-life associated with the terminal slope Lambda (z) of the semi logarithmic drug concentration-time curve, calculated as 0.693/Lambda (z).
Total Apparent Clearance (CL/F) of Midazolam | Predose, 0.5, 1, 1.5, 2, 3 , 4, 6, 8, 10, 12, 16, 24, 30, 36 and 48 hours postdose on Day 1 during Treatment A and on Day 7 during Treatment B
  The CL/F is defined as Dose/AUC (0-infinity).
Total Apparent Clearance (CL/F) of 1-Hydroxymidazolam | Predose, 0.5, 1, 1.5, 2, 3 , 4, 6, 8, 10, 12, 16, 24, 30, 36 and 48 hours postdose on Day 1 during Treatment A and on Day 7 during Treatment B
  The CL/F is defined as Dose/AUC (0-infinity).
Total Apparent Clearance (CL/F) of Warfarin | Predose, 0.5, 1, 2 , 4, 6, 9, 12, 16, 24, 36, 48, 72, 96, 120, 144 and 168 hours postdose on Day 3 during Treatment A and on Day 9 during Treatment B
  The CL/F is defined as Dose/AUC (0-infinity).
Apparent Volume of Distribution (Vd/F) of Midazolam | Predose, 0.5, 1, 1.5, 2, 3 , 4, 6, 8, 10, 12, 16, 24, 30, 36 and 48 hours postdose on Day 1 during Treatment A and on Day 7 during Treatment B
  The Vd/F is defined as Dose/[Lambda (z)*AUC (0-infinity)].
Apparent Volume of Distribution (Vd/F) of 1-Hydroxymidazolam | Predose, 0.5, 1, 1.5, 2, 3 , 4, 6, 8, 10, 12, 16, 24, 30, 36 and 48 hours postdose on Day 1 during Treatment A and on Day 7 during Treatment B
  The Vd/F is defined as Dose/[Lambda (z)*AUC (0-infinity)].
Apparent Volume of Distribution (Vd/F) of Warfarin | Predose, 0.5, 1, 2 , 4, 6, 9, 12, 16, 24, 36, 48, 72, 96, 120, 144 and 168 hours postdose on Day 3 during Treatment A and on Day 9 during Treatment B
  The Vd/F is defined as Dose/[Lambda (z)*AUC (0-infinity)].
Maximum Observed Effect (Emax) for Prothrombin Time (PT) | Predose, 2 , 6, 12, 16, 24, 30, 36, 40, 48, 54, 60, 66, 72, 96, 120, 144 and 168 hours postdose on Day 3 during Treatment A and on Day 9 during Treatment B
  The Emax for prothrombin time (PT) will be assessed.
Maximum Observed Effect (Emax) for activated Partial Thromboplastin Time (aPTT) | Predose, 2 , 6, 12, 16, 24, 30, 36, 40, 48, 54, 60, 66, 72, 96, 120, 144 and 168 hours postdose on Day 3 during Treatment A and on Day 9 during Treatment B
  The Emax for activated partial thromboplastin time (aPTT) will be assessed.
Maximum Observed Effect (Emax) for International Normalized Ratio (INR) | Predose, 2 , 6, 12, 16, 24, 30, 36, 40, 48, 54, 60, 66, 72, 96, 120, 144 and 168 hours postdose on Day 3 during Treatment A and on Day 9 during Treatment B
  The Emax for international normalized ratio (INR) will be assessed.
Time to Reach the Maximum Plasma Concentration (Tmax) of JNJ-42847922 | 2 hours postdose on Day 1 to Day 6; 2 and 26 hours postdose on Day 7; 2 hours postdose on Day 9 during Treatment B
  The Tmax is the time to reach the maximum observed plasma concentration of JNJ-42847922.
Area Under the Plasma Concentration-Time Curve From 0 to 168 Hours (AUC[0-168]) Post Dose of Warfarin | Predose, 0.5, 1, 2 , 4, 6, 9, 12, 16, 24, 36, 48, 72, 96, 120, 144 and 168 hours postdose on Day 3 during Treatment A and on Day 9 during Treatment B
  The AUC(0-168hrs) is the area under the plasma concentration-time curve from 0 to 168 hours post dosing.
Area Under the Plasma Concentration-Time Curve From 0 to 168 Hours (AUC[0-168]) Post Dose of JNJ-42847922 | 2 hours postdose on Day 1 to Day 6; 2 and 26 hours postdose on Day 7; 2 hours postdose on Day 9 during Treatment B
  The AUC(0-168hrs) is the area under the plasma concentration-time curve from 0 to 168 hours post dosing.
Pharmacodynamic Effect by Using Bond and Lader Visual Analogue Scale (B and L VAS) | Day -1 of Treatment A dosing
  The B and L VAS will be performed to measure effects of a JNJ-42847922 on the duration of the pharmacodynamic effect of midazolam. The B and L VAS includes 16 questions with VAS scales to rate subjective feelings.
Pharmacodynamic Effect by Using Bond and Lader Visual Analogue Scale (B and L VAS) | 4 hours postdose on Day 1 during Treatment A
  The B and L VAS will be performed to measure effects of a JNJ-42847922 on the duration of the pharmacodynamic effect of midazolam. The B and L VAS includes 16 questions with VAS scales to rate subjective feelings.
Pharmacodynamic Effect by Using Bond and Lader Visual Analogue Scale (B and L VAS) | 8 hours postdose on Day 1 during Treatment A
  The B and L VAS will be performed to measure effects of a JNJ-42847922 on the duration of the pharmacodynamic effect of midazolam. The B and L VAS includes 16 questions with VAS scales to rate subjective feelings.
Pharmacodynamic Effect by Using Bond and Lader Visual Analogue Scale (B and L VAS) | Day -1 of Treatment B dosing
  The B and L VAS will be performed to measure effects of a JNJ-42847922 on the duration of the pharmacodynamic effect of midazolam. The B and L VAS includes 16 questions with VAS scales to rate subjective feelings.
Pharmacodynamic Effect by Using Bond and Lader Visual Analogue Scale (B and L VAS) | 4 hours postdose on Day 7 during Treatment B
  The B and L VAS will be performed to measure effects of a JNJ-42847922 on the duration of the pharmacodynamic effect of midazolam. The B and L VAS includes 16 questions with VAS scales to rate subjective feelings.
Pharmacodynamic Effect by Using Bond and Lader Visual Analogue Scale (B and L VAS) | 8 hours postdose on Day 7 during Treatment B
  The B and L VAS will be performed to measure effects of a JNJ-42847922 on the duration of the pharmacodynamic effect of midazolam. The B and L VAS includes 16 questions with VAS scales to rate subjective feelings.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious AEs | Screening up to follow-up visit (7 to 14 days after last study procedure)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Overland Park, Kansas, United States